CLINICAL TRIAL: NCT07129772
Title: A Multicenter, Single Arm Phase II Study on Pembrolizumab and Chemotherapy as Perioperative Treatment Followed by Nasopharyngectomy and Maintenance Pembrolizumab for Locally Recurrent Nasopharyngeal Carcinoma (PINNACLE)
Brief Title: Perioperative Chemotherapy and Immunotherapy for Locally Recurrent Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Sun Yat-sen University (Other); Changhua Christian Hospital (Other); National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PINNACLE
Record Dates: First submitted 2025-08-11; First posted 2025-08-19 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-07

CONDITIONS: Nasopharyngeal Cancer Recurrent; Nasopharyngeal Cancinoma (NPC)
Keywords: Nasopharyngeal carcinoma; Locally recurrent; Perioperative treatment; Immune checkpoint inhibitor; Chemotherapy; Minimally invasive surgery
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Gemcitabine; Cisplatin; pembrolizumab; Single Person

STUDY DESIGN:
Intervention Model Description: Perioperative chemotherapy and immune checkpoint inhibitor for locally recurrent nasopharyngeal carcinoma
Masking Description: Inapplicable
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perioperative chemotherapy and immune checkpoint inhibitor for recurrent nasopharyngeal carcinoma (Experimental): Perioperative chemotherapy and immune checkpoint inhibitor every 3 weeks for up to 6 cycles followed by radically minimally invasive surgery e.g. endoscopic nasopharyngectomy or transoral robotic-assisted nasopharyngectomy and maintenance pembrolizumab for a total of 1 year for locally recurrent nasopharyngeal carcinoma.
  Interventions: Drug: Gemcitabine (GEM); Drug: Cisplatin; Drug: PEMBROLIZUMAB (alone or when added to a regimen above)

INTERVENTIONS:
Drug: Gemcitabine (GEM) — Gemcitabine, cisplatin and pembrolizumab for up to 6 cycles followed by minimally invasive surgery (either endoscopic nasopharyngectomy or transoral robotic-assisted nasopharyngectomy) and maintenance pembrolizumab for a total of 1 year for locally recurrent nasopharyngeal carcinoma
  Other Names: Gemcitabine
Drug: Cisplatin — Gemcitabine, cisplatin and pembrolizumab for up to 6 cycles followed by minimally invasive surgery (either endoscopic nasopharyngectomy or transoral robotic-assisted nasopharyngectomy) and maintenance pembrolizumab for a total of 1 year for locally recurrent nasopharyngeal carcinoma
Drug: PEMBROLIZUMAB (alone or when added to a regimen above) — Gemcitabine, cisplatin and pembrolizumab for up to 6 cycles followed by minimally invasive surgery (either endoscopic nasopharyngectomy or transoral robotic-assisted nasopharyngectomy) and maintenance pembrolizumab for a total of 1 year for locally recurrent nasopharyngeal carcinoma
  Other Names: Keytruda

SUMMARY:
Nasopharyngeal carcinoma (NPC) is an endemic malignancy in Southern China and southeast Asia. Despite intensive radical therapy, between 15% and 30% of NPC patients develop relapse. Recent phase III randomized-controlled trials conducted in China demonstrated an improvement of progression-free survival with combinational therapy immune checkpoint inhibitors (ICI) (camrelizumab, toripalimab, and tislelizumab, respective) and chemotherapy gemcitabine (G) and cisplatin (P) compared with chemotherapy GP alone for recurrent or metastatic NPC. However, none of these studies have described in details the treatment outcomes of those subjects with locally recurrent NPC only, and whether any of these patients would undergo radical surgery to remove the residual locally recurrent NPC after ICI and chemotherapy. Continuation of the same ICI as maintenance therapy may only be the treatment option for these patients who were recruited into these phase III trials, unless if they withdrew from the study and opted for radical resection. While continuing the same ICI may still lead to persistent objective response and disease control, there is a possibility of tumor recurrence leading to unresectable disease and a worse survival outcome, or unexpected, rare but recognized immune-related emergent adverse events with ICI. Radical resection after maximal response to ICI and chemotherapy for patients with locally recurrent NPC only may provide a chance of cure of the disease and these patients may be obviated from continuous exposure to ICI therapy.

In view of the above, we are now proposing a phase II single-arm study on perioperative pembrolizumab and chemotherapy followed by radical surgery for locally recurrent NPC. As a collateral study, we will also perform single-cell DNA and RNA sequencing and proteomics study to observe the tumor and immune microenvironment which certainly helps us decipher the mechanisms of tumor response at genomic, transcriptomic and proteomic levels.

DETAILED DESCRIPTION:
This is a multi-centre single-arm phase II study on perioperative treatment with pembrolizumab and chemotherapy GP for 6 cycles followed by radical surgery and maintenance pembrolizumab for another 11 cycles (up to 17 cycles of pembrolizumab in total).

All eligible patients shall receive preoperative treatment with pembrolizumab at 200mg fixed dose, with chemotherapy G: 1000-1250mg/m2 on day 1 and day 8 and P: 80-100mg/m2 on day 1 (or carboplatin AUC=5 on day 1 replacing cisplatin at the treating physician's discretion), given every 3 weeks for 6 cycles followed by radical surgery (open or minimally invasive surgery) at the discretion of treating surgeons, and subsequently maintenance pembrolizumab for another 11 cycles (up to 17 cycles of pembrolizumab for 1 year).

All recruited patients will undergo reassesment imaging scans after 3 and 6 cycles of pembrolizumab and chemotherapy GP. They will then undergo radical surgery within 4 to 6 weeks of the 6th cycle of pembrolizumab and chemotherapy GP. Subsequently, within 4 to 6 weeks of radical surgery, they will continue the remaining 11 cycles of pembrolizumab 200mg fixed dose every 3 weeks up to 17 cycles in total.

Magnetic resonance imaging (MRI) of the head and neck and positron emission tomography with integrated computed tomography (PET-CT) scan will be performed at baseline before study intervention and after 3 and 6 cycles of pembrolizumab and chemotherapy GP and before radical surgery, to evaluate tumor response. After radical surgery, all recruited subjects will undergo repeat MRI and contrast-enhanced computed tomography (CT) scan of the thorax and abdomen every 3 months during the 1st year, then every 4 months during the 2nd year, every 6 months during the 3rd and 4th year, and yearly from the 5th year onwards.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of histologically confirmed locally recurrent (rT2-T4, N0-N1, M0) NPC (undifferentiated carcinoma with Epstein-Barr virus (EBV) infection by either presence of Epstein-Barr virus encoded RNA (EBER) in in-situ hybridization of the recently obtained tumor specimen before study entry) or an elevation of plasma EBV DNA in the subject's peripheral blood), staged according to the 8th edition of American Joint Committee on Cancer/Union for International Cancer Control (AJCC/UICC) staging classification (TNM-8). All patients should NOT have received any form of anti-tumor treatment for their locally recurrent NPC before joining the study. However, prior radical treatment for their NPC at diagnosis is allowed if there is at least a 6-month interval between prior radical treatment and the start of study intervention of this study.
2. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
3. Aged ≥18 years old
4. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
5. All eligible patients must be magnetic resonance imaging of T1, T2 and T1-contrast enhanced sequences of the head and neck region and PET-CT scan within 30 days of study entry.
6. Modified Charlson Comorbidity Score <2
7. Adult Comorbidity Evaluation (ACE)-27 Index <2
8. Pre-existing peripheral neuropathy <=1
9. Have adequate organ function as defined in the following table (Table 5.1.1).
10. Body Weight >30kg
11. For women of childbearing potential, a negative serum or urine pregnancy test within 14 days prior to the start of treatment for their NPC. Women will be considered postmenopausal if they are amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply: - Women 1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
12. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
13. Must have a life expectancy of at least 12 weeks.

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment or 5 half-lives, whichever is shorter.
2. Has a diagnosis of severe active scleroderma, lupus, other rheumatologic or autoimmune disease within the past 3 months before study recruitment. Patients with a documented history of clinically severe autoimmune disease or a syndrome requiring systemic steroids or immunosuppressive agents will not be allowed on this study. Subjects with vitiligo or resolved childhood asthma/atopy are an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections are not excluded from the study. Subjects with hypothyroidism stable on hormone replacement are not excluded from this study.
3. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
4. Has had any prior monoclonal antibody before study entry, including but not limited to anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another costimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137 etc).
5. Has had prior chemotherapy or targeted small molecule therapy (including sorafenib or other anti-vascular endothelial growth factor inhibitor) before study entry. Patients who received radical radiation therapy and chemotherapy (but not immune checkpoint inhibitors or any form of immunotherapy) for their previously untreated nasopharyngeal carcinoma at diagnosis was allowed to join this study, provided that such radical treatment was completed >6 months before study entry.
6. Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded. Other exceptions may be considered with Sponsor consultation.

   Note: Participants with low risk early-stage prostate cancer defined as below are not excluded: Stage T1c or T2a with a Gleason score ≤6 and a prostate-specific antigen (≤10 ng/ml) either treated with definitive intent or untreated in active surveillance that has been stable for the past year prior to study allocation.
7. Has known carcinomatous meningitis (also known as leptomeningeal carcinomatosis).
8. Has an active infection requiring intravenous systemic therapy or hospital admission.
9. Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
10. Has a history or current evidence of any condition, therapy, or laboratory abnormality, including psychiatric or substance abuse disorder, that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
11. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 31 weeks after the last dose of trial treatment.
12. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies). Routine checking for Anti-HIV1 or Anti-HIV2 is not mandatory.
13. Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (HCV; defined as HCV RNA [qualitative] is detected) infection.
14. Has received a live vaccine 30 days prior to the first dose of trial treatment.
15. Has experienced Grade 4 toxicity on treatment with prior radiation.
16. Has experienced Grade 3-4 intracranial toxicity (hypophysitis or central nervous system toxicity) with either prior intracranial radiation and/or chemotherapy.
17. Is taking > 4mg/day of dexamethasone or its equivalent at the start of immunotherapy or has required > 4mg/day of dexamethasone or its equivalent for 3 consecutive days within 1 week of starting treatment.
18. Allergies and adverse drug reaction to the following: History of allergy to study drug components; History of severe hypersensitivity reaction to any monoclonal antibody.
19. Any unresolved toxicity National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade >=2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria. (a) Patients with Grade >=2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician. (b) Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with pembrolizumab may be included only after consultation with the Study Physician.
20. Major surgical procedure (as defined by the Investigator within 28 days prior to the first dose of IP. Local surgery of isolated lesions for palliative intent is acceptable.
21. History of allogenic organ transplantation.
22. History of leptomeningeal carcinomatosis.
23. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) >=470ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart).
24. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) >=470ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart).
25. Current or prior use of immunosuppressive medication within 14 days before the first dose of pembrolizumab. The following are exceptions to this criterion: (a) Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection) (b) Systemic corticosteroids at physiologic doses not to exceed <> of prednisone or its equivalent (c) Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | 36 months
  Rate of the absence of all detectable cancer cells in tissue samples examined under a microscope by certified pathologists after perioperative treatment with gemcitabine, cisplatin and pembrolizumab and minimally invasive surgery (either endoscopic nasopharyngectomy or transoral robotic-assisted nasopharyngectomy) for locally recurrent nasopharyngeal carcinoma

SECONDARY OUTCOMES:
Objective response rate | 36 months
  Rate of objective response as per RECIST 1.1 or irRECIST
Major pathological response | 36 months
  Rate of the less than or equal to 10% of detectable and viable cancer cells in tissue samples examined under a microscope by certified pathologists after perioperative treatment with gemcitabine, cisplatin and pembrolizumab and minimally invasive surgery (either endoscopic nasopharyngectomy or transoral robotic-assisted nasopharyngectomy) for locally recurrent nasopharyngeal carcinoma
Recurrence-free survival | 36 months
  Rate of survival calculated from the time of the date of written informed consent to the date of radiologically confirmed recurrence of nasopharyngeal carcinoma or the date of death from any cause
Overall survival | 36 months
  Rate of survival calculated from the time of the date of written informed consent to the date of death from any cause
Toxicity profiles | 36 months
  Number of participants who suffer from adverse events or serious adverse events according to Common Terminology Criteria for Adverse Events version 5.0
Biomarkers | 36 months
  Number of participants found to have biomarkers including tumor and blood biomarkers predictive of objective response to perioperative treatment with gemcitabine, cisplatin and pembrolizumab

CONTACTS AND LOCATIONS:
Overall Officials: Victor Ho-Fun Lee, MD, Principal Investigator — Department of Clinical Oncology, The University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Individual patient data of this study will not be shared unless a request with an approved research proposal is submitted to the principal investigator for consideration.

REFERENCES:
- [Background] Chan ATC, Lee VHF, Hong RL, Ahn MJ, Chong WQ, Kim SB, Ho GF, Caguioa PB, Ngamphaiboon N, Ho C, Aziz MASA, Ng QS, Yen CJ, Soparattanapaisarn N, Ngan RK, Kho SK, Tiambeng MLA, Yun T, Sriuranpong V, Algazi AP, Cheng A, Massarelli E, Swaby RF, Saraf S, Yuan J, Siu LL. Pembrolizumab monotherapy versus chemotherapy in platinum-pretreated, recurrent or metastatic nasopharyngeal cancer (KEYNOTE-122): an open-label, randomized, phase III trial. Ann Oncol. 2023 Mar;34(3):251-261. doi: 10.1016/j.annonc.2022.12.007. Epub 2022 Dec 16. PMID 36535566